CLINICAL TRIAL: NCT00000241
Title: Flupenthixol Decanoate in Methamphetamine Smoking
Brief Title: Flupenthixol Decanoate in Methamphetamine Smoking - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Friends Research Institute, Inc. (Other)
Purpose: Treatment
Other Study IDs: NIDA-07200-1; R01-07200-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: methamphetamine dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Flupenthixol

INTERVENTIONS:
Drug: Flupenthixol

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of flupenthixol decanoate for treatment of methamphetamine dependence. Also, study will compare flupenthixol with desipramine in blocking methamphetamine self-administration.

ELIGIBILITY:
Please contact site for information.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58
Dates: Start 1994-02; Study Completion 1996-05

PRIMARY OUTCOMES:
Methamphetamine use

CONTACTS AND LOCATIONS:
Overall Officials: Frank Gawin, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States